CLINICAL TRIAL: NCT00390923
Title: Testing a Full Substitution Therapy Approach As Treatment of Tobacco Dependence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary results did not support the utility of combining selegeline + NRT.
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Tobacco Control Research Initiative (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, MD, PhD, CCFP, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 170/2006
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Nicotine Dependence
Keywords: smoking; nicotine dependence; double-blind; placebo-controlled; randomized; full substitution therapy; selegiline
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Selegiline; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Selegiline + nicotine replacement therapy
- 2 (Placebo Comparator)
  Interventions: Drug: placebo + nicotine replacement therapy

INTERVENTIONS:
Drug: Selegiline + nicotine replacement therapy — Participants will begin selegiline once a day during Week 1, and dose will be graduated to full study dosage (10 mg/day) by adding an evening intake (a.m. and p.m. dosing) for Weeks 2-8. Day 15 of the trial represents target quit day and the transdermal nicotine patch (21 mg/24hr) will be applied at this time. Patches will be worn in conjunction with study medication for Weeks 3-8, after which the patch will be removed and study medication tapered throughout Week 9.
  Arms: 1
Drug: placebo + nicotine replacement therapy — Participants will begin placebo once a day during Week 1, and dose will be graduated to full study dosage (10 mg/day) by adding an evening intake (a.m. and p.m. dosing) for Weeks 2-8. Day 15 of the trial represents target quit day and the transdermal nicotine patch (21 mg/24hr) will be applied at this time. Patches will be worn in conjunction with study medication for Weeks 3-8, after which the patch will be removed and study medication tapered throughout Week 9.
  Arms: 2

SUMMARY:
This study will test a new medication strategy designed to help smokers quit. It will combine selegiline, a drug currently approved and available for the treatment of Parkinson's disease, with a nicotine skin patch. Forty nicotine-dependent smokers will enrolled in this study. Twenty will receive placebo (inactive pill) plus nicotine patch, and twenty will receive selegiline plus nicotine patch. Once enrolled in the study, subjects will visit the Nicotine Dependence Clinic at CAMH on a weekly basis for assessment of smoking behavior, a brief health check, collection of breath and urine samples (necessary to drug levels and nicotine levels), and receive brief individual counseling designed to help them stop smoking. The medication phase of this study lasts 9 weeks. A follow-up visit will be conducted six months after trial completion. At that point, health and behavioral measures will be re-assessed.

DETAILED DESCRIPTION:
This pilot study utilizes a double-blind, two-armed design to evaluate the efficacy of combining oral selegiline with transdermal nicotine patch for smoking cessation in 40 nicotine-dependent smokers. After successful completion of 3 screening visits (to ensure medical and psychiatric eligibility criteria are met), subjects will be randomized into one of two experimental groups:

1. selegiline (10 mg/day) + NRT (21 mg/24 hr)
2. matching placebo + NRT (21 mg/24 hr)

Randomization will be performed through the use a random number list to generate 50% selegiline/50% placebo and also 50% male/50% female within each of those treatment groups.

Participants will begin selegiline (or placebo) once a day during Week 1, and dose will be graduated to full study dosage (10 mg/day) by adding an evening intake (a.m. and p.m. dosing) for Weeks 2-8. Day 15 of the trial represents target quit day and the transdermal nicotine patch (21 mg/24hr) will be applied at this time. Patches will be worn in conjunction with study medication for Weeks 3-8, after which the patch will be removed and study medication tapered throughout Week 9.

Subjects will present weekly to the Nicotine Dependence Clinic where they will provide breath, urine and blood samples as required, receive brief smoking cessation counseling and complete questionnaires regarding their smoking behavior and psychological state. A post-trial physical will be conducted upon completion of Week 9. Monthly follow-up phone interviews will be conducted for 5 months and subjects will be re-assessed in the NDC for a 6-month follow-up.

Trial Objectives

1. To determine if combination of selegiline hydrochloride and NRT (full substitution to tobacco) is superior to NRT alone + placebo (partial substitution) for smoking cessation in nicotine dependent smokers.

   * The primary hypothesis is that full substitution (selegiline + NRT) will be superior to placebo + NRT for achievement of 7-day point prevalence smoking abstinence rates at the end of trial abstinence rates (Day 49-56) assessment in nicotine-dependent cigarette smokers.
   * Secondary hypothesis 1a is that full substitution (selegiline + NRT) will be superior to NRT for achievement of last four weeks of trial (Days 29-56) smoking abstinence rates in nicotine-dependent cigarette smokers.
   * Secondary hypothesis 1b is that full substitution (selegiline + NRT) will be superior to NRT for achievement 6-month post target quit date smoking abstinence rates in nicotine-dependent cigarette smokers.
2. To determine if treatment retention and study medication compliance will be higher in the full substitution (selegiline + NRT) group as compared to the NRT group during the 8-week smoking cessation trial.

   Hypothesis 2 is that treatment retention and study medication compliance will be higher in the full substitution (selegiline + NRT) group as compared to the NRT group during the 8-week smoking cessation trial.
3. To determine if full substitution (selegiline + NRT) reduces nicotine craving and withdrawal symptoms as compared to NRT group during the 8-week smoking cessation trial.

   Hypothesis 3 is that full substitution treatment will lead to significant reductions in tobacco withdrawal and craving ratings compared to NRT group.
4. To determine adverse events profile in nicotine-dependent smokers of the combination of selegiline and NRT as compared to NRT.

Hypothesis 4 is that selegiline in combination with NRT will be well-tolerated and that rates of adverse events will not be significantly different between subjects assigned to full substitution as compared to NRT group.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for nicotine dependence with FTND score > 5.
* Smoke at least 15 cigarettes (3/4 pack) daily (averaged over 1 week, in the past 1 month).
* At the time of initial evaluation, are motivated to quit smoking in the next 30 days.
* Have made at least one unsuccessful attempt to quit smoking in the past year.
* At baseline, have expired breath CO level > 10.
* Are between ages 18-70 years old.
* Weigh at least 100 lbs (45.5 kg, selegiline dose < 0.22 mg/kg).
* No previous use of nicotine replacement products in the one month prior to randomization.
* Have the capacity to give informed consent, and are English-speaking.

Exclusion Criteria:

* Have present or past diagnoses of schizophrenia, bipolar disorder, PTSD, BPD or major depressive illness.
* Have abused alcohol or other drugs of abuse (cocaine, opiates, benzodiazepines, etc) in 6 months prior to randomization into the trial (based on clinical evaluation including self-report, and confirmed by positive urine).
* Demonstrate serious medical conditions (i.e. abnormal liver function [as evidenced by AST, ALT or bilirubin values 2x ULN], unstable cardiovascular disease, significant blood abnormalities).
* Exhibit or have history of clinical hypertension.
* Exhibit active peptic ulcer disease.
* Are pregnant, are trying to become pregnant, or are currently breastfeeding.
* Are on current medication regimes that include antidepressants, or sympathomimetic agents, or meperidine and other meperidine-opioids which may have interactions with selegiline.
* Known hypersensitivity to selegiline or NRT.
* Are from the same household as another study participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Seven-day point prevalence smoking abstinence at end of trial (abstinence based on self-reported smoking abstinence verified by CO levels < 10 ppm) | 9 weeks

SECONDARY OUTCOMES:
Last four weeks of Trial Continuous smoking abstinence rates (verified by CO < 10 ppm) | 4 weeks
Seven-day point prevalence smoking abstinence | end of treatment, six-month follow-up
Treatment retention (based on survival analysis and number of weeks a subject completes in the trial) | upon completion
Time line follow back for cigarettes smoked, alcohol and caffeinated beverage use | Weeks 1-8; six-month follow-up
Tobacco craving as assessed by Tiffany scale for smoking urges | Weeks 1, 4 and 8; 6-month follow-up
DSM-IV nicotine withdrawal symptom checklist | Weeks 1, 4 and 8; 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Henningfield JE, Goldberg SR. Nicotine as a reinforcer in human subjects and laboratory animals. Pharmacol Biochem Behav. 1983 Dec;19(6):989-92. doi: 10.1016/0091-3057(83)90405-7. PMID 6657732
- [Background] Stolerman IP, Shoaib M. The neurobiology of tobacco addiction. Trends Pharmacol Sci. 1991 Dec;12(12):467-73. doi: 10.1016/0165-6147(91)90638-9. PMID 1792691
- [Background] Caggiula AR, Donny EC, White AR, Chaudhri N, Booth S, Gharib MA, Hoffman A, Perkins KA, Sved AF. Cue dependency of nicotine self-administration and smoking. Pharmacol Biochem Behav. 2001 Dec;70(4):515-30. doi: 10.1016/s0091-3057(01)00676-1. PMID 11796151
- [Background] Fowler JS, Volkow ND, Wang GJ, Pappas N, Logan J, Shea C, Alexoff D, MacGregor RR, Schlyer DJ, Zezulkova I, Wolf AP. Brain monoamine oxidase A inhibition in cigarette smokers. Proc Natl Acad Sci U S A. 1996 Nov 26;93(24):14065-9. doi: 10.1073/pnas.93.24.14065. PMID 8943061
- [Background] Robinson TE, Berridge KC. The neural basis of drug craving: an incentive-sensitization theory of addiction. Brain Res Brain Res Rev. 1993 Sep-Dec;18(3):247-91. doi: 10.1016/0165-0173(93)90013-p. PMID 8401595
- [Background] Robinson TE, Berridge KC. Incentive-sensitization and addiction. Addiction. 2001 Jan;96(1):103-14. doi: 10.1046/j.1360-0443.2001.9611038.x. PMID 11177523
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961